CLINICAL TRIAL: NCT03883373
Title: Comparison Between Alveolar Bone Graft With Only Cancellous Bone, and Alveolar Bone Graft With Cancellous Bone Combined With Nasal Cavity Floor's Reconstruction Using a Cortical Block
Brief Title: Alveolar Bone Graft Cortical Nasal Floor
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL19_0136
Record Dates: First submitted 2019-03-18; First posted 2019-03-20 (Actual); Last update posted 2019-08-12 (Actual); Status verified 2019-03

CONDITIONS: Alveolar Cleft Operated on an Alveolar Bone Graft
Keywords: alveolar graft; cancellous bone; cortical block; nasal floor
MeSH Terms: interventions — Alveolar Bone Grafting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cortical group: Group of patient who had an alveolar bone graft with cancellous bone and a cortical block
  Interventions: Procedure: alveolar bone graft with cancellous bone and a cortical block
- Cancellous group: Group of patient who had an alveolar bone graft with cancellous bone only
  Interventions: Procedure: alveolar bone graft with cancellous bone only

INTERVENTIONS:
Procedure: alveolar bone graft with cancellous bone and a cortical block — alveolar bone graft with cancellous bone only
  Groups: Cortical group
Procedure: alveolar bone graft with cancellous bone only — alveolar bone graft with cancellous bone only
  Groups: Cancellous group

SUMMARY:
Alveolar bone graft is one of the main step of the surgical care of the patients who are suffering from cleft lip and palate. They are usually performed before the lateral incisor eruption, at about 5 years old and using cancellous bone taken from the iliac crest.

The aim of the study is to show if adding a cortical graft to the cancellous cause more complications, which may be source of partial or total graft loss in the 6 month following the observation

DETAILED DESCRIPTION:
This is an observational, retrospective and monocentric study. To be included, patients had to suffer from a clef lip and palate or alveolar cleft and had to have an alveolar bone graft with gingivo-periosteoplasty in the pediatric plastic surgery unit of the Montpellier hospital from June 1999 to Mai 2016. They were divided into two groups : the first with patients who had a cortical and cancellous bone graft and the second with patients who had a cancellous graft only.

Both groups were followed 6 mounts after the operation to look for the occurence of complications which lead to a graft loss. Bilateral cleft are seen as 2 graft events

ELIGIBILITY:
Inclusion criteria:

* Patients with a clef lip and palate or alveolar cleft
* Grafted in the Montpellier pediatric surgery unit from june 1999 to mai 2016
* Followed during 6 months of post operative follow up

Exclusion criteria:

* No post operative follow up
* other alveolar bone graft in the past medical history

Ages: 3 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Patients who are suffering from clef lip and palate or alveolar cleft and had to have an alveolar bone graft with gingivo-periostoplasty in the pediatric plastic surgery unit of the Montpellier hospital from June 1999 to Mai 2016
Sampling Method: Non-Probability Sample
Enrollment: 302 (Actual)
Dates: Start 1999-06-01 (Actual); Primary Completion 2016-05-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Complication events | 6 months
  Analyze retrospective of the electronic medical record was made as followed: read of peri-operative and post-operative reports, looking for complications during the 6 months of post operative follow up
  Analyze of the electronic medical record was made as followed: read of peri-operative and post-operative reports, looking for readmission in Pediatric Emergency department and finally read of the report of the clinical control 1 month after the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CAPTIER, MD.PhD, Study Director — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France